CLINICAL TRIAL: NCT03663673
Title: Comparison of Two Different Skin Creams and Their Effect on Transepidermal Water Loss (TEWL) in Pediatric and Adult Patients With Atopic Dermatitis: A Pilot Study
Brief Title: Effect of Different Skin Creams on TEWL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: End Allergies Together (EAT) (Unknown)
Responsible Party: Principal Investigator, Sayantani B. Sindher, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNP 47028
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis; emollient; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis | interventions — EpiCeram

STUDY DESIGN:
Intervention Model Description: Prospective, single center, clinical pilot study to test the hypothesis that lipid rich EpiCeram® is superior in improving skin barrier function compared to Aveeno Daily Moisturising Sheer Hydration Lotion®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Clinical pilot study (Other): To compare skin barrier function, assessed by TEWL AUC, between non-lesional areas of the skin treated with EpiCeram®, Aveeno Daily Moisturising Sheer Hydration Lotion®, and no emollient use over a period of one week.
  Interventions: Drug: EpiCeram; Drug: Aveeno Daily Moisturising Sheer Hydration Lotion®

INTERVENTIONS:
Drug: EpiCeram — To compare skin barrier function, assessed by TEWL AUC, between non-lesional areas of the skin treated with EpiCeram®, Aveeno Daily Moisturising Sheer Hydration Lotion®, and no emollient use over a period of one week.
Drug: Aveeno Daily Moisturising Sheer Hydration Lotion® — To compare skin barrier function, assessed by TEWL AUC, between non-lesional areas of the skin treated with EpiCeram®, Aveeno Daily Moisturising Sheer Hydration Lotion®, and no emollient use over a period of one week.

SUMMARY:
Prospective, single center, clinical pilot study to test the hypothesis that lipid rich EpiCeram® is superior in improving skin barrier function compared to Aveeno Daily Moisturising Sheer Hydration Lotion®.

DETAILED DESCRIPTION:
Prospective, single center, clinical pilot study to test the hypothesis that lipid rich EpiCeram® is superior in improving skin barrier function compared to Aveeno Daily Moisturising Sheer Hydration Lotion®.

Primary Objective: To compare skin barrier function, assessed by TEWL AUC, between non-lesional areas of the skin treated with EpiCeram®, Aveeno Daily Moisturising Sheer Hydration Lotion® or no emollient use for one week.

Secondary Objectives: To assess lipid and protein profiles of skin tape strips from non-lesional skin, after a week of either EpiCeram®, Aveeno Daily Moisturising Sheer Hydration Lotion® or no treatment.

Exploratory Objectives :

* To study whether the effects on TEWL on lesional and non-lesional skin persist 24 hours after cessation of therapy.
* To evaluate whether baseline food and environmental allergy sensitization (assessed via skin prick testing during screening) affects the outcomes. See protocol section 3.1 for allergen details.
* A central repository of blood samples will be stored for future use to assess plasma biomarkers to help characterize clinical outcome data.

ELIGIBILITY:
Inclusion Criteria:

1. Parent guardian must be able to understand and provide informed consent per Institutional Review Board (IRB) guidelines and regulations.
2. Male or female participants, between the ages of 0 to 40 years will be included
3. Diagnosis of moderate to severe active AD (Scoring Atopic Dermatitis (SCORAD) score > 26) without a history or current manifestations of eczema herpeticum (EH)
4. AD affecting at least 3 different skin areas (contralateral arms and one lower extremity)

Exclusion Criteria:

1. Inability or unwillingness of a parent guardian to give written informed consent, or to comply with study protocol.
2. Participants with skin disease other than AD that might compromise the stratum corneum barriers (e.g., bullous diseases, psoriasis, cutaneous T-cell lymphoma (also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease).
3. Known or suspected immunosuppression
4. Severe concomitant illness(es)
5. History of serious life-threatening reaction to latex, tape, or adhesives
6. Has received total body phototherapy (e.g., ultraviolet light B [UVB], psoralen ultraviolet light A [PUVA], tanning beds [>1 visit per week]) within 30 days of the Enrollment Visit
7. Use of topical corticosteroids, topical immunomodulatory agents (such as calcineural inhibitors and crisaborole), or topical antibiotics on the upper or lower extremities within 7 days of the Enrollment Visit
8. Has taken a bleach bath within 7 days of the Enrollment Visit
9. Use of systemic antibiotics, antiparasitics, antivirals, or antifungals within 7 days of the Enrollment Visit.

Ages: 1 Day to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Skin barrier function | 2 weeks
  Skin barrier function, assessed by TEWL

SECONDARY OUTCOMES:
Baseline food and environmental allergy sensitization | 2 weeks
  Skin prick testing

CONTACTS AND LOCATIONS:
Overall Officials: Sayantani Sindher, M.D., Principal Investigator — Stanford Health Care; Kari Nadeau, M.D., PhD, Study Chair — Stanford Health Care
Locations (1):
- Sean N Parker Center For Allergy and Asthma Research, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No